CLINICAL TRIAL: NCT03850145
Title: Evaluation of the Efficacy of an Educational Program Through Video Conference
Brief Title: Educational Program Through Video Conference for Inhaled Therapies in Cystic Fibrosis Patients
Acronym: Visio-Respir
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0054
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
Keywords: inhaled therapy; physiotherapist; educational program
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Educational programs are essential for cystic fibrosis patients who need to take several different drugs every day. Compliance is often klow in these patients, and clinicals and paramedics try to increase it, through educational programs. As for inhaled therapies, the CF center of Montpellier uses a video conference tool to educate patients. The program may involve either the physiotherapist or the doctor or both. Through the present study, the investigators would like to evaluate the current practice at the CF center of Montpellier and verify if patients feel that the physiotherapist could handle the program on his own, without the support of a physician.

ELIGIBILITY:
Inclusion criteria:

* CF patients
* patient regularly assessed at the CF center of Montpellier
* major patients
* patients who recently enrolled a video conference educational program or who will soon be part of it

Exclusion criteria:

* patients not able to participate to a video conference educational program, due to lack of tools at their home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CF patients consulting at the CF center of Montpellier (France)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
acceptability of the therapeutic education program by videoconference | 1 day
  acceptability of the therapeutic education program by videoconference with a satisfaction questionnaire
need for the presence of the referring physician in relation to a session of therapeutic education carried out by the physiotherapist alone | 1 day
  need for the presence of the referring physician in relation to a session of therapeutic education carried out by the physiotherapist alone with a satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Davide CAIMMI, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided